CLINICAL TRIAL: NCT07306936
Title: Computer Guided Single Needle Arthrocentesis With Platelets Rich Plasma Injection in the Management of Temporomandibular Joint Internal Derangement
Brief Title: Computer Guided Single Needle Arthrocentesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-12-25-RE-Shepared
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorder (TMD); Internal Derangement; Anterior Disc Displacement
Keywords: temporomandibular disorder; intra-articular injection; internal derangement; anterior disc displacement; computer-assisted; Computer-aided design; computer-aided manufacturing; software; shepard cannula
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with TMJ ID + reduction managed with computer-guided single needle arthrocentesis (Experimental): Patients with TMJ ID + reduction managed with computer-guided single needle arthrocentesis in adjunct to PRP intra-articular injection.
  Interventions: Device: Computer-guided single needle arthrocentesis
- Patients with TMJ ID + reduction managed with conventional free hand single needle arthrocentesis (Placebo Comparator): Patients with TMJ ID + reduction managed with conventional free hand single needle arthrocentesis in adjunct to PRP intra-articular injection
  Interventions: Device: conventional free hand single needle arthrocentesis

INTERVENTIONS:
Device: Computer-guided single needle arthrocentesis — Patients with TMJ ID + reduction managed with computer-guided single needle arthrocentesis in adjunct to PRP intra-articular injection
  Arms: Patients with TMJ ID + reduction managed with computer-guided single needle arthrocentesis
Device: conventional free hand single needle arthrocentesis — Patients with TMJ ID + reduction managed with conventional free hand single needle arthrocentesis in adjunct to PRP intra-articular injection.
  Arms: Patients with TMJ ID + reduction managed with conventional free hand single needle arthrocentesis

SUMMARY:
The intra-articular injection is considered the first line of minimally invasive treatment in temporomandibular joint with internal derangement (TMJ-ID) patients who do not respond to conservative treatment. The single-needle technique arthrocentesis has emerged to add reliability, convenience, ease the performance of the procedure, and eliminate the need for multiple punctures the Aim of this study is to assess clinical applicability and therapeutic outcomes of computer guided single needle arthrocentesis with platelet rich plasma using Shepard's cannula, in comparison with conventional free-hand technique, in the management of disc displacement with reduction of the TMJ.

DETAILED DESCRIPTION:
A total of 24 patients with a magnetic resonance imaging (MRI) diagnosis of reducing disc displacement will be included and assigned randomly into one of two groups. Computer-guided arthrocentesis with PRP will be performed on patients in the study group using the single needle technique by Shepard cannula technique; while the conventional free hand technique will be performed in the control group. Procedure-related parameters will be assessed, while Clinical evaluation will be conducted on day 1, 1 and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with internal derangement according to Wilkes stage I and II.
2. Adult patients above 18 years old.
3. Patients who would not respond to conservative treatment as a first line of treatment

Exclusion Criteria:

1. Patients with Wilkes stage III, IV, V.
2. Patients suffering from any systemic diseases, platelets function disorders, fibrinogen deficiency.
3. History of mandibular fracture.
4. Lactating, pregnant or planning pregnancy women.
5. Patients receiving anticoagulation treatment or NSAIDS within 48 hours preoperatively, corticosteroid injection at treatment site within 1 month or systemic use of corticosteroids within 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
objective assessment of joint function and mandibular excursion | 3 months
  Clinical evaluation will be based on the Helkimo's clinical dysfunction index (Di), which is a part of the Helkimo index that provides an objective assesment of joint function and mandibular excursion.
  All patients will be assessed immediately post-operative, 1 and 3 months. Postoperative clinical evaluation values will be compared to the preoperative baseline preoperative values.

SECONDARY OUTCOMES:
Duration of the Operation | intraoperative
  Total procedural time consumed starting from the application of topical antiseptic up to the end of the procedure will be measured and compared between both groups. In the Computer-Guided group, the time for needle injection will be further computed to determine the actual injection time in the procedure bar from the guide installation time and patient preparation.

CONTACTS AND LOCATIONS:
Overall Officials: yehia El-Mahallawy, Phd, Principal Investigator — Faculty of Dentistry, Alexandria University, Alexandria, Alexandria
Locations (1):
- Outpatient clinics of Faculty of Dentistry, Alexandria University, Egypt Alexandria, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study